CLINICAL TRIAL: NCT04712383
Title: Impact of Wearable Health Devices and Health and Wellness Behavior Change Support on Health Outcomes and Healthcare Costs
Brief Title: Impact of Wearable Health Devices and Wellness Behavior Change Support on Health Outcomes and Healthcare Costs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Fitbit LLC (Industry); Massachusetts eHealth Initiative (Unknown)
Responsible Party: Principal Investigator, Steven Bird, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H00021669; 2020 - MeHI - 01 (Other Grant/Funding Number: Massachusetts eHealth Initiative)
Record Dates: First submitted 2021-01-11; First posted 2021-01-15 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Health Behavior
Keywords: health behavior; fitness
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fitbit Care intervention arm (Experimental): The experimental arm will receive the full Fitbit Care product suite (Fitbit wrist-worn device, Fitbit connected weight scale, and Fitbit Premium + Health Coaching service). Participants in the experimental arm will also be offered support in improving health behaviors that are important to them, including activity, nutrition, sleep, stress management, and medication adherence.
  Interventions: Combination Product: Fitbit Care intervention arm
- Fitbit study control arm (No Intervention): Participants in the control arm will have access to standard healthcare benefits available to all employees, but will not have access to any of the Fitbit Care interventions

INTERVENTIONS:
Combination Product: Fitbit Care intervention arm — Entire suite of Fitbit Care.
  Arms: Fitbit Care intervention arm

SUMMARY:
The purpose of this study is to measure the impact of consumer-grade wearable health devices and behavior change support services, including health coaching, on health behaviors, biometrics, and healthcare costs. The study will be a randomized controlled trial with 700 participants who are employees of UMass Memorial Health Care in which 350 participants (control group) receive standard wellness and medical benefits and services for UMass Memorial Health Care employees and in which 350 participants (intervention group) receive these same standard benefits and services as well as the full Fitbit Care product suite (Fitbit wrist-worn device, Fitbit connected weight scale, and Fitbit Premium + Health Coaching service). Participants in the intervention group will be offered support in improving health behaviors that are important to them, including activity, nutrition, sleep, stress management, and medication adherence. They will also be offered support in tying these behaviors to their health goals, including blood pressure management, blood sugar management, cholesterol management, weight loss, smoking cessation, etc.

The hypothesis is that those employees in the intervention group will experience improved results compared to those in the control group. It is believed that they will have improved health behaviors, improved biometrics, and lower total healthcare costs (fewer complications, fewer hospitalizations, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Employed by UMassMemorial Health Care
* Receive benefits from UMassMemorial Health Care
* Have a smartphone

Exclusion Criteria:

* Pregnant
* Unable to consent
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Change in total medical expenditures for calendar year 2020 to 2021 | 12 months
  Change in total medical expenditures from calendar year 2020 to 2021 Participant insurance claim information will be analyzed to determine the change in total medical expenditures from 2020 to 2021 and the results will be compared between the intervention and control groups.
Changes in Biometric Outcomes | 12 months
  Participants will have biometric screening including body weight at the beginning and end of the study that will be used to determine the change in that biometric over the course of the study, and the results will be compared between the intervention and control groups.
Changes in Biometric Outcomes | 12 months
  Participants will have biometric screenings including waist circumference at the beginning and end of the study that will be used to determine the change in that biometric over the course of the study, and the results will be compared between the intervention and control groups.
Changes in Biometric Outcomes | 12 months
  Participants will have biometric screenings including blood pressure at the beginning and end of the study that will be used to determine the change in that biometric over the course of the study, and the results will be compared between the intervention and control groups.
Changes in Biometric Outcomes | 12 months
  Participants will have biometric screenings including LDL cholesteral at the beginning and end of the study that will be used to determine the change in that biometric over the course of the study, and the results will be compared between the intervention and control groups.
Changes in Biometric Outcomes | 12 months
  Participants will have biometric screenings including HDL cholesteral at the beginning and end of the study that will be used to determine the change in that biometric over the course of the study, and the results will be compared between the intervention and control groups.
Changes in Biometric Outcomes | 12 months
  Participants will have biometric screenings including hemoglobin A1c at the beginning and end of the study that will be used to determine the change in that biometric over the course of the study, and the results will be compared between the intervention and control groups.
Changes in self-reported health behaviors and levels of motivation and confidence in making improvements | 3 months, 6 months, 9 months, and 12 months
  Participants will complete a health behavior survey (addresses overall health, nutrition, activity, sleep, mindfulness, alcohol, and smoking behaviors as well as levels of motivation and confidence in making improvements) at the beginning of the study and every three months until the end of the study. This will be used to determine changes in behaviors, motivation, and confidence over the course of the study, and the results will be compared between the intervention and control groups. This is not done via a scale, but answers range from Strongly agree, to Somewhat agree, to Neither agree nor disagree, to Somewhat disagree, to Strongly disagree.

SECONDARY OUTCOMES:
Proportion of participants achieving target biometric outcomes | 12 months
  Participants will have biometric screenings (including body weight, waist circumference, blood pressure, hemoglobin A1c, and LDL and HDL cholesterol) at the beginning and end of the study that will be used to determine, for each biometric, the percentage of participants in each study arm who reach standard clinical target values, and the percentage of participants will be compared between the intervention and control groups.
Proportion of participants achieving categorical improvement in biometric outcomes | 12 months
  Participants will have biometric screenings (including body weight, waist circumference, blood pressure, hemoglobin A1c, and LDL and HDL cholesterol) at the beginning and end of the study that will be used to determine, for each biometric, the percentage of participants in each study arm who improve at least one clinical category (for example, from stage 2 hypertension to stage 1 hypertension, and the percentage of participants will be compared between the intervention and control groups.
Correlations between responses to health behavior survey and total medical expenditure and biometric outcomes | 12 months
  Participant responses to the health behavior survey (behaviors as well as levels of motivation and confidence in making improvements) will be analyzed for correlations with changes in total medical expenditures and biometric outcomes.
Changes in metrics collected by Fitbit devices and Fitbit app | weekly and totaled over 12 months
  For participants in the intervention group, changes in steps taking collected by Fitbit devices and in the Fitbit app will be analyzed over the course of the study.
Changes in metrics collected by Fitbit devices and Fitbit app | weekly and totaled over 12 months
  For participants in the intervention group, changes in active zone minutes collected by Fitbit devices and in the Fitbit app will be analyzed over the course of the study.
Changes in metrics collected by Fitbit devices and Fitbit app | weekly and totaled over 12 months
  For participants in the intervention group, changes in hours of sleep collected by Fitbit devices and in the Fitbit app will be analyzed over the course of the study.
Correlations between metrics collected by Fitbit devices and Fitbit app and total medical expenditure and biometric outcomes | 12 months
  For participants in the intervention group, changes in metrics collected by Fitbit devices and in the Fitbit app will be analyzed for correlations with changes in total medical expenditures and biometric outcomes.
Correlations between engagement with health coach and total medical expenditure and biometric outcomes | 12 months
  For participants in the intervention group, engagement with the health coach in the Fitbit app will be measured based on the number of text messages and interactions with the health coaching action plan and analyzed for correlations with changes in total medical expenditures and biometric outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Bird, MD, Principal Investigator — UMass Memorial Healthcare
Locations (1):
- UMassMemorial Health Care, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
IPD is not planned to share with other researchers.

REFERENCES:
- [Derived] Howard-Wilson S, Ching J, Gentile S, Ho M, Garcia A, Ayturk D, Lazar P, Hammerquist N, McManus D, Barton B, Bird S, Moore J, Soni A. Efficacy of a Multimodal Digital Behavior Change Intervention on Lifestyle Behavior, Cardiometabolic Biomarkers, and Medical Expenditure: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Oct 30;13:e50378. doi: 10.2196/50378. PMID 39475852